CLINICAL TRIAL: NCT00835640
Title: A Relative Bioavailability Study of 180 mg Fexofenadine Hydrochloride Tablets Under Fed Conditions.
Brief Title: Fexofenadine Hydrochloride 180 mg Tablets Under Non-Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: R01-862
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Results first posted 2009-08-04 (Estimated); Last update posted 2009-08-20 (Estimated); Status verified 2009-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — fexofenadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Fexofenadine 180 mg tablets
- 2 (Active Comparator)
  Interventions: Drug: ALLEGRA® 180 mg tablets

INTERVENTIONS:
Drug: Fexofenadine 180 mg tablets — 1 x 180 mg
  Arms: 1
Drug: ALLEGRA® 180 mg tablets — 1 x 180 mg
  Arms: 2

SUMMARY:
This study will compare the relative bioavailability (rate and extent of absorption) of 180 mg Fexofenadine Hydrochloride tablets manufactured for TEVA Pharmaceuticals Industries, Ltd. with that of 180 mg ALLEGRA® Tablets by Aventis Pharmaceuticals, Inc. following a single oral dose (1 x 180 mg tablet) in healthy adult volunteers under fed conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* All volunteers selected for this study will be healthy, non-smoking men and women 18 to 55 years of age, inclusive, at the time of dosing. The volunteer's body mass index (BMI) is less that or equal to 30.
* If female and :

  * Of child bearing potential, is practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence; or
  * Is postmenopausal for at least 1 year; or
  * Is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).

Exclusion Criteria:

* Volunteers with a recent history of drug or alcohol addiction or abuse.
* Volunteers with the presence of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease (as determined by the clinical investigators).
* Volunteers whose clinical laboratory test values are outside the accepted reference range and when confirmed on re-examination are deemed to be clinically significant.
* Volunteers demonstration a positive hepatitis B surface antigen screen, hepatitis C antibody screen or a reactive HIV antibody screen.
* Volunteers demonstrating a positive drug abuse screen when screened for this study.
* Female volunteers who are currently breast feeding.
* Female volunteers who are demonstrating a positive pregnancy screen.
* Volunteers with a history of allergic response(s) to fexofenadine or related drugs.
* Volunteers with a history of clinically significant allergies including drug allergies.
* Volunteers with a clinically significant illness during the 4 weeks prior to Period I dosing (as determined by the clinical investigators).
* Volunteers who currently use or reports using tobacco or nicotine-containing products within 90 days prior to Period I dosing.
* Volunteers who have taken any drug known to induce or inhibit hepatic drug metabolism in the 30 days prior to Period I dosing.
* Volunteers who report donating greater than 150 mL of blood within 30 days prior to Period I dosing. All subjects will by advised not to donate blood for four weeks after completing the study.
* Volunteers who have donated plasma (e.g. plasmapheresis) within 14 days prior to Period I dosing. All subjects will be advised not to donate plasma for four weeks after completing the study.
* Volunteers who report receiving any investigational drug within 30 days prior to Period I dosing.
* Volunteers who report taking any prescription medication in the 14 days prior to Period I dosing, with the exception of topical products without systemic absorption.
* Volunteers who have been on an abnormal diet during the 28 days prior to Period I dosing.
* Volunteers who report an intolerance of direct venipuncture.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2002-01; Primary Completion 2002-01 (Actual); Study Completion 2002-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D Carlson, Pharm. D., Principal Investigator — PRACS Institute, Ltd.
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Fexofenadine Hydrochloride First: 180 mg Fexofenadine Hydrochloride Tablets test product dosed in first period followed by 180 mg Allegra® Tablets reference product dosed in the second period.
- Allegra® First: 180 mg Allegra® Tablets reference product dosed in first period followed by 180 mg Fexofenadine Hydrochloride Tablets test product dosed in the second period.
Period: First Intervention
Arm/Group | Fexofenadine Hydrochloride First | Allegra® First
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Washout of 7 Days
Arm/Group | Fexofenadine Hydrochloride First | Allegra® First
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Fexofenadine Hydrochloride First | Allegra® First
Started | 12 | 12
Completed | 11 | 12
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fexofenadine Hydrochloride First | Allegra® First | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 8 | 9 | 17
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian | 0 | 1 | 1
  White | 12 | 11 | 23
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Cmax = Maximum Observed Concentration.
Description: Bioequivalence based on Cmax.
Time Frame: Blood samples collected over a 48 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Fexofenadine Hydrochloride: 180 mg Fexofenadine Hydrochloride Tablets test product dosed in either period.
- Allegra®: 180 mg Allegra® Tablets reference product dosed in either period.
Arm/Group | Fexofenadine Hydrochloride | Allegra®
Number analyzed (Participants) | 23 | 23
ng/mL | 311.45 (99.83) | 382.48 (119.07)
Statistical Analysis 1: Comparison: Fexofenadine Hydrochloride vs Allegra®; Test type: Non-Inferiority or Equivalence — The ANOVA model was utilized in comparing the effects between the test and reference products. Differences were declared statistically significant at the 5% level (p<0.05); Ratio of the T/R geometric mean x 100 = 81.33 — To establish bioequivalence, the ratio of the mean must fall within 80-125

2. Primary Outcome: AUC0-t = Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration (Per Participant)
Description: Bioequivalence based on AUC0-t.
Time Frame: Blood samples collected over a 48 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Fexofenadine Hydrochloride | Allegra®
Number analyzed (Participants) | 23 | 23
ng*h/mL | 1894.48 (562) | 2159.85 (671.03)
Statistical Analysis 1: Comparison: Fexofenadine Hydrochloride vs Allegra®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 87.87 — To establish bioequivalence, the ratio of the mean must fall within 80-125

3. Primary Outcome: AUC0-inf = Area Under the Concentration-time Curve From Time Zero to Infinity.
Description: Bioequivalence based on AUC0-inf.
Time Frame: Blood samples collected over a 48 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Fexofenadine Hydrochloride | Allegra®
Number analyzed (Participants) | 23 | 23
ng*h/mL | 2061.26 (627.94) | 2324.97 (718.31)
Statistical Analysis 1: Comparison: Fexofenadine Hydrochloride vs Allegra®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 88.45 — To establish bioequivalence, the ratio of the mean must fall within 80-125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator is not permitted to discuss or publish trial results.